CLINICAL TRIAL: NCT01475136
Title: A Single Dose Pharmacokinetic Study of LY2140023 in Subjects With Hepatic Impairment
Brief Title: A Study of LY2140023 in Hepatically-Impaired Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12677; H8Y-MC-HBCH (Other: Eli Lilly and Company); 2011-003033-34 (EudraCT Number)
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2013-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — LY 2140023

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2140023 (Experimental): A single oral dose of 80 milligrams (mg) LY2140023 administered on Day 1.
  Interventions: Drug: LY2140023

INTERVENTIONS:
Drug: LY2140023

SUMMARY:
This study will explore how liver impairment affects blood levels of LY2140023 (a prodrug) and its active metabolite (LY404039).

DETAILED DESCRIPTION:
The study included 4 groups, based on the Child-Pugh classification of hepatic impairment as follows:

Group 1: Participants with normal hepatic function (Control); Group 2: Participants with mild hepatic impairment (Child-Pugh class A); Group 3: Participants with moderate hepatic impairment (Child-Pugh class B); and Group 4: Participants with severe hepatic impairment (Child-Pugh class C).

ELIGIBILITY:
Inclusion Criteria:

* Male participants agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023
* Female participants of child-bearing potential who test negative for pregnancy at screening and agree to use a reliable method of birth control for the duration of the study and for at least 3 months after the last dose of LY2140023
* Female participants who are postmenopausal. Postmenopausal is defined as no menses for at least 1 year, or a plasma follicle stimulating hormone (FSH) value of greater than 40 units per liter (IU/L), unless the participant is taking hormone replacement therapy
* Have a body mass index (BMI) between 19 and 40 kilograms per square meter (kg/m^2), inclusive at the time of screening
* Have clinical laboratory test results within the normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have sitting blood pressure and heart rate compatible with their disease state, as determined by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site
* Control participants that have normal hepatic function, as determined by medical history and physical examination
* Hepatically-impaired participants that have stable hepatic impairment (for example, alcoholic, posthepatitis, biliary cirrhosis, or cryptogenic) classified as Child-Pugh class A, B, or C (mild, moderate, or severe impairment) who are considered acceptable for participation in the study by the investigator

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 90 days from last dosing of an investigational product (other than the investigational product used in this study); or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2140023, LY404039, related compounds, or any components of the formulation
* Have previously discontinued after receiving at least 1 dose of LY2140023 or completed this study or any other study investigating LY2140023 and or LY404039
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption (except cholecystectomy), metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have evidence of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, or depression)
* Participants who answer 'yes' to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the Columbia Suicide Severity Rating Scale (C-SSRS), or answer "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior) on the "Suicidal Behavior" portion of the C-SSRS; and the ideation or behavior occurred within the past 3 months
* Have increased risk of seizures based on a history of:

  * One or more seizures (except for a single simple febrile seizure [lacking focality and lasting less than 15 minutes, not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * Head trauma with loss of consciousness or a post-concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * CNS infection, uncontrolled migraine or transient ischemic attack (TIA) within 1 year; stroke with persistent neurological deficit (focal or diffuse). Uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning. TIA is defined as "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * Brain surgery
  * Electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, sharp-slow wave complexes, or as locally defined)
  * Brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (does not include hydrocephalus unless treated by shunt or resulting in neurological deficits)
* Known substance dependence unless approved prescription medication such as opiates, or known regular use of drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Women who are pregnant or intend to get pregnant during the study or within 3 months after the last dose of investigational product
* Women who are breast feeding or lactating
* Have donated blood of more than 500 milliliters (mL) within the last 3 months prior to the screening
* Are organ transplant participants or have taken immunosuppressants following any organ transplant
* Have shown signs of variceal bleeding during the last 2 months prior to screening (except for participants with severe hepatic impairment, detailed in exclusion criterion)
* Show evidence of irritable bowel syndrome or chronic diarrhea
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), and are participants unwilling to stop alcohol consumption for 96 hours predose until after 48 hours post-dose (1 unit equals 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Have a clinically significant abnormality in the neurological examination
* Participants judged prior to dosing to be at suicidal risk by the investigator
* Participants who are unwilling to refrain from smoking from midnight prior to dosing until 6 hours postdose or are unable to abide by the Clinical Research Unit (CRU) restrictions
* Are on total parenteral nutrition (TPN)
* Take oral anticoagulants for therapeutic use
* Exhibit any other condition, which, in the opinion of the investigator would preclude participation in the study
* Show evidence of pruritus or skin exfoliation
* Have an eosinophil count >1.5 x 10^9/liter (L)
* Have electrolyte imbalance alerts (clinically significant changes in calcium magnesium, or sodium)
* Control Participants:

  * Have any medically significant history of neurologic disease, cancer, or cardiac, respiratory, metabolic, hepatic, renal, gastrointestinal (except appendectomy), dermatological, venereal, hematological disorder or disease
  * Have creatinine clearance (CrCl) less than 80 milliliters per minute (mL/min), as calculated by the Cockcroft-Gault equation:

Men: [(140 - age) x (weight in kilograms [kg])] / [72 x (serum creatinine in mg/100 mL)]; or [(140 - age) x (weight in kg)] / [0.81 x (serum creatinine in micromoles per liter [μmol/L])] Women in both of the above equations: (x 0.85)

* Show evidence of significant active neuropsychiatric disease in the opinion of the investigator
* Evidence of hepatitis B and/or positive hepatitis B surface antigen (HBsAg)
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Intend to use over-the-counter medication (including herbal remedies/health supplements) within 7 days prior to dosing, or prescription medication (other than hormone replacement therapy as described above) within 14 days prior to dosing

  * Mild Hepatic Impaired Participants (Child-Pugh A):
* show evidence of any significant active disease other than that responsible for or associated with hepatic impairment
* have a platelet count of less than 50 x 10^9 cells/L, unless after consultation with the Lilly Clinical Pharmacologist (CP), they are considered as acceptable for participation in the study

  * Moderate and Severe Hepatic Impaired Participants (Child-Pugh B and C):
* Show evidence of any significant active disease other than that responsible for or associated with moderate or severe hepatic impairment
* Have shown signs of spontaneous bacterial peritonitis within 6 months prior to dosing
* Have severe hyponatremia
* Show evidence of significant active neuropsychiatric disease
* Have hepatic encephalopathy (Grades 2 to 4)
* Have hemoglobin concentrations <9.0 grams per deciliter (g/dL)
* Show signs of hepatocellular carcinoma
* Have a surgical portosystemic shunt
* Have a platelet count of less than 40 x 10^9 cells/L (moderate impairment) or less than 30 x 10^9 cells/L (severe impairment), unless after consultation with the Lilly CP they are considered as acceptable for participation in the study
* Have shown signs of variceal bleeding during the last 2 weeks prior to screening (severe hepatic impaired participants only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred, Hungary

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (Pts) were enrolled in Group 3 (moderate hepatic impairment) after satisfactory interim safety and pharmacokinetic (PK) data was obtained from ≥3 Pts in Group 2 (mild hepatic impairment). Pts were enrolled in Group 4 (severe hepatic impairment) after satisfactory interim safety and PK data was obtained from ≥3 Pts in Group 3.
Groups:
- LY2140023-Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of 80 milligrams (mg) LY2140023 on Day 1.
- LY2140023-Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of 80 mg LY2140023 on Day 1.
- LY2140023-Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of 80 mg LY2140023 on Day 1.
- LY2140023-Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of 80 mg LY2140023on Day 1.
Period: Overall Study
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment
Started | 7 | 9 | 9 | 12
Received 1 Dose of Study Drug | 7 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 7
Not Completed | 1 | 3 | 3 | 5
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- LY2140023-Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of 80 mg LY2140023 on Day 1.
- Total: Total of all reporting groups
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment | Total
Number analyzed (Participants) | 7 | 9 | 9 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (2.5) | 57.4 (5.9) | 56.8 (4.0) | 53.9 (7.3) | 56.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 5 | 18
  Male | 3 | 6 | 3 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 9 | 9 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 9 | 9 | 12 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 4 | 2 | 5 | 12 | 23
  Germany | 3 | 7 | 4 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve (AUC) of LY2140023 and LY404039
Description: LY404039 is the active metabolite of LY2140023. AUC from zero to infinity AUC(0-∞) is presented.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, and 48 hours postdose
Population: All participants who received 1 dose of LY2140023, did not have an incidence of vomiting within 5 hours postdose, and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment
Number analyzed (Participants) | 5 | 6 | 6 | 5
nanograms*hours per milliliter (ng*h/mL)
  LY2140023 | 1420 (34) | 1360 (30) | 836 (57) | 926 (22)
  LY404039 | 2710 (16) | 3290 (28) | 2570 (28) | 2640 (33)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of LY2140023 and LY404039
Description: LY404039 is the active metabolite of LY2140023.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, and 48 hours postdose
Population: All participants who received 1 dose of LY2140023, did not have an incidence of vomiting within 5 hours postdose, and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment
Number analyzed (Participants) | 5 | 6 | 6 | 5
nanograms/milliliter (ng/mL)
  LY2140023 | 332 (27) | 305 (29) | 211 (41) | 194 (25)
  LY404039 | 440 (10) | 517 (23) | 431 (28) | 403 (28)

3. Primary Outcome: Pharmacokinetics: Time of Maximal Concentration (Tmax) of LY2140023 and LY404039
Description: LY404039 is the active metabolite of LY2140023.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, and 48 hours postdose
Population: All participants who received 1 dose of LY2140023, did not have an incidence of vomiting within 5 hours postdose, and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment
Number analyzed (Participants) | 5 | 6 | 6 | 5
hours
  LY2140023 | 3.00 [2.00 to 4.00] | 2.50 [2.00 to 3.00] | 2.50 [1.00 to 4.00] | 2.00 [2.00 to 3.00]
  LY404039 | 4.00 [3.00 to 4.00] | 4.00 [3.00 to 4.00] | 3.50 [2.00 to 4.00] | 4.00 [3.00 to 4.00]

ADVERSE EVENTS:
Arm/Group | LY2140023-Normal Hepatic Function | LY2140023-Mild Hepatic Impairment | LY2140023-Moderate Hepatic Impairment | LY2140023-Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 5/7 | 5/6 | 4/6 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2140023-Normal Hepatic Function (N=7) | LY2140023-Mild Hepatic Impairment (N=6) | LY2140023-Moderate Hepatic Impairment (N=6) | LY2140023-Severe Hepatic Impairment (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days